CLINICAL TRIAL: NCT03007810
Title: An Ascending Single Dose Study of the Pharmacokinetics, Safety and Tolerability of Hemay005 in Healthy Male Subjects
Brief Title: Safety and Pharmacokinetics of Hemay005 In Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Bio-Tech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM005PS1S01
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemay005 (Experimental): Four subjects in cohort 1 and six subjects in each cohort (2 to 6) will receive Hemay005.
  Interventions: Drug: Hemay005
- Placebo (Placebo Comparator): Two subjects in each cohort (cohorts 2 to 6) will receive placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Hemay005 — Subjects will be randomized into 6 cohorts(10mg, 20mg, 40mg, 80mg, 120mg, 180mg) orally single dose
  Arms: Hemay005
Drug: Placebos — Subjects will be randomized into 5 cohorts(20mg, 40mg, 80mg, 120mg, 180mg) orally single dose
  Arms: Placebo

SUMMARY:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis. This study is the first administration of Hemay005 in humans to establish the initial safety, tolerability, and pharmacokinetic profile following single doses of Hemay005. A total of approximately 44 subjects will be randomized into 6 cohorts(10mg, 20mg, 40mg, 80mg, 120mg, 180mg), approximately 8 healthy subjects will be enrolled (6 active and 2 placebo) at each dose cohort by sentinel method(1 active and 1 placebo,5 active and 1 placebo), with the exception of 10mg (4 active) cohort. This study includes an 28-day Screening Period, a 1-day Treatment Period, and an End of Study Visit occurring approximately 11days (±3 days) after study drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18 to 60 years;
2. Bodyweight（BW）≥ 50kg, Body mass index (BMI) in 18-28 (including upper and lower limit of the range);
3. All male subjects must agree and commit to the use of a reliable contraceptive regimen(including vasoligation, abstinence, using a condom) for the duration of the study(from screening until 6 months after the last dose);
4. Ability to understand and be willing to sign a written informed consent before study entry;
5. Subjects would have good communication with the investigator and could comply with protocol.

Exclusion Criteria:

1. A history of clinically severe gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or haematological disorders;
2. Have a known history of hypersensitivity to any medicine or food, or allergy to the test article or any of the excipient of the test article;
3. Have a gastrointestinal, hepatic or renal condition that may influence drug absorption or metabolism;
4. A history of chronic infection (ie, tuberculosis);
5. A medical history of any clinically significant medical disease or surgery within 4 weeks of the screening;
6. Clinically significant laboratory abnormal results at screening or prior to the first dose of study drug;
7. Clinically significant abnormal 12-lead ECG or vital signs ( systolic pressure <90 mmHg or >140 mmHg, diastolic pressure <50 mmHg or >90 mmHg; radial pulse rate <50 bpm or >100 bpm);
8. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening;
9. Recent history of frequent alcohol consumption, defined by average intake of greater than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol content, or 150 mL wine), Participants who are unable to abstain from smoking during the study or quitting smoking for less than 3 months;
10. Positive urine screen for drug and cigarettes, positive breath test for alcohol;
11. Subjects who use soft drugs (ie marijuana )within 3 months of the screening and entire study duration or hard drugs (ie cocaine, phencyclidine ) within 1 year of the screening and entire study duration;
12. Dietary habits or food intolerances which will interfere with the requirements for participants to consume a standardised diet whilst confined to the clinical unit;
13. Participants who eat special food (Including grapefruit and/or Xanthine diet) for 14 days prior to dosing or any caffeine containing food or drinks, i.e. chocolate for 48 hours prior to dosing or drinking alcohol for 24 hours prior to dosing and not will stop to intake above food and drinks;
14. Use of any drug that inhibits or induces hepatic metabolism of drugs within 30 days of planned study drug administration and entire study duration (e.g. inducers: barbiturates, carbamazepine, rifampicin, phenytoin, glucocorticoid and omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones and antihistamines);
15. Participant who received any medicine within 14 days of the initial dose of study drug;
16. Have received other clinical trials treatment within 3 months prior to study;
17. Participants who have donated of blood (>400 mL) within 4 weeks of the study, or plan to donate of blood during of the study and 4 weeks after the study;
18. Subjects cannot complete the study due to other reasons or by the investigator's judgment

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | Day 1 up to Day 11±3

SECONDARY OUTCOMES:
Cmax | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Maximum observed plasma concentration
Tmax | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Time of maximum concentration
AUCt | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
AUC∞ | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
t1/2 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Terminal elimination half-life
CL/F | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Apparent total plasma clearance
Vz/F | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 hours post-dose
  Apparent total volume of distribution
Cumulative urinary excretion | pre-dose, 0-4 hours，4-8 hours，8-12 hours，12-24 hours，24-36 hours，36-48 hours post-dose
Accumulative urine excretion rate | pre-dose, 0-4 hours，4-8 hours，8-12 hours，12-24 hours，24-36 hours，36-48 hours post-dose
Renal clearance | pre-dose, 0-4 hours，4-8 hours，8-12 hours，12-24 hours，24-36 hours，36-48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No